CLINICAL TRIAL: NCT04995939
Title: Evaluation of the Effects of Preoperative Neutrophil/Lymphocyte Ratio, Albumin Level, and Various Risk Scorings on Postoperative Pulmonary Complications in Thoracic Surgery. Prospective Observational Study
Brief Title: Preoperative Laboratory Parameters and Scorings Systems on Postoperative Pulmonary Complications in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulay Ulger, Principal investigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2230
Record Dates: First submitted 2021-07-09; First posted 2021-08-09 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2021-11

CONDITIONS: Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laboratory parameters and Scoring systems — Neutrophil/ Lymphocite ratio, albumin level and scoring systems has been evaluated.

SUMMARY:
Postoperative pulmonary complications (PPC) emerge as a major risk that determines the morbidity and mortality of patients after surgery. PPCs affect the length of hospital stay and increase health costs. Because of this reason, it is important to predict PPCs before surgery. There are many studies on scoring systems that can be effective in predicting PPCs. The most frequently used ones are the Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) risk index, the Nutritional Risk Score (NRS), and the American Society of Anesthesiologist (ASA) score. ARISCAT risk index is mostly evaluated in operations performed other than thoracic surgery. Since the thoracic wall, mediastinum or lungs are directly intervened in thoracic surgery operations, the expected PPCs in these patients may be different from those expected in other surgical groups. Therefore, the ARISCAT risk index may be insufficient to evaluate PPCs in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective thoracotomy or video assisted thoracic surgery with general anesthesia
* BMI < 35 kg/m2
* Age 18 - 75 years old
* Expected operative time more than 60 minutes

Exclusion Criteria:

* History of lung surgery
* Advanced lung-heart disease
* Having a previous COVID-19 pneumonia

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-75 years who are scheduled for elective thoracotomy or VATS, who have not had previous thoracic surgery, and without advanced lung and heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Distribution of patients who developed one or more postoperative pulmonary complications according to preoperative neutrophil/lymphocyte ratio, albumin value, ARISCAT risk index, nutritional risk score, and ASA physical status. | Time to preoperative visit and through study completion, an average of three months.
  1. Effectiveness of the ARISCAT risk scoring index [ Time Frame: postoperative first 30 days ]
     to investigate the effectiveness of the ARISCAT risk scoring index in predicting the development of PPC in patients undergoing thoracic surgery.
  2. Correlation between ASA physical status (1-3) and PPC [ Time Frame: postoperative first 30 days ]
  3. Correlation between NRS ( nutritional risk score) score (0-3) and PPC [ Time Frame: postoperative first 30 days ]
  4. Correlation between preoperative albumin values (gram / dl) and PPC [ Time Frame: postoperative first 30 days ]
  5. Correlation between preoperative neutrophil/lymphocyte ratio and PPC [ Time Frame: postoperative first 30 days ]

SECONDARY OUTCOMES:
Distribution of patients who developed one or more postoperative pulmonary complications according to age, gender, BMI and preoperative SpO2 level. | Time to preoperative visit and up to 30 days.
  1. Correlation between age (years) and PPC [ Time Frame: postoperative first 30 days
  2. Correlation between gender(male or female) and PPC [ Time Frame: postoperative first 30 days ]
  3. Correlation between BMI (kg/m^2) and PPC [ Time Frame: postoperative first 30 days ]
  4. Correlation between Preoperative Sp02(>96%, 91%-95%, <90%) and PPC [ Time Frame: postoperative first 30 days ]

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Chest Diseases and Chest Surgery Training and Research Hospital, Ankara, Keçioören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulger G, Sazak H, Baldemir R, Zengin M, Kaybal O, Incekara F, Alagoz A. The effectiveness of ARISCAT Risk Index, other scoring systems, and parameters in predicting pulmonary complications after thoracic surgery. Medicine (Baltimore). 2022 Jul 29;101(30):e29723. doi: 10.1097/MD.0000000000029723. PMID 35905198